CLINICAL TRIAL: NCT03533842
Title: Interactive Care Assessment of Risk Factors and Emergency Levels
Brief Title: Validation of a Computerized Triage Algorithm for Ophthalmic Emergencies
Acronym: iCare
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MGJ_2017_29
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Emergencies
Keywords: Triage; Algorithms; Emergencies; Eyes emergencies; Ophtalmology
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
The investigators conceived a computerized interactive tool for Emergency Triage, based on a patient's symptoms, medical history and background. Using this tool, the patient (alone or helped by a nurse / supporting person) presenting to an ophthalmologic ER, should be able to detect and prioritize his most urgent symptoms (A,B), in opposition to less urgent (C) or non urgent symptoms (D). To test the validity of this tool, each patient presenting at the Rothschild Foundation ER (Paris, France) with an ophthalmological problem should be included and sorted by the algorithm before the medical consultation. Neither the patient nor the practitioner are aware of the scoring (A,B,C,D) defined by the algorithm. The practitioner should then give his own emergency scoring (A,B,C,D) after patient examination. A total of 1000 patients is expected.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the Emergency Room for Ophthalmologic concerns

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seeking an emergency consultation at the Ophthalmologic emergency unit
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Comparison between the emergency level defined by iCare and the emergency level decided by the physician at the end of his consultation (gold standard). | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Guedj, Principal Investigator — Institut Arthur Vernes
Locations (2):
- France (2):
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Instutut Arthur Vernes, Paris